CLINICAL TRIAL: NCT00952133
Title: Randomized Double Blind Study to Evaluate the Efficacy of IV Palo w/ IV Dexamethasone vs IV Palo for Prevention of Immediate & Delayed Post-Operative Nausea/Vomiting in Subj Undergoing Laparoscopic Surgeries w/a High Emetogenic Risk
Brief Title: Efficacy of IV Palo With IV Dexamethasone vs IV Palo for Prevention of Immediate & Delayed PONV
Acronym: PONV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: H08-605
Record Dates: First submitted 2009-07-30; First posted 2009-08-04 (Estimated); Results first posted 2014-03-31 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-03

CONDITIONS: PONV
Keywords: PONV; Outpatient surgery; Laparoscopic abdominal surgery; Laparoscopic gynecologic surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Palonosetron; Saline Solution; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palonosetron with Dexamethasone (Experimental): Women/Men 18-55 scheduled for surgery 1-3 hours in duration will be given .075 mg IV Palonosetron (Aloxi) with 8mg IV Dexamethasone (Decadron) before surgery.
  Interventions: Drug: Palonosetron with Dexamethasone
- Palonosetron only (Placebo Comparator): Women/Men 18-55 scheduled for surgery 1-3 hours in duration will be given .075 mg IV Intravenous Palonosetron and Saline solution
  Interventions: Drug: Palonosetron only

INTERVENTIONS:
Drug: Palonosetron only — The placebo arm will be given a dose of IV palonosetron only, and saline solution prior to surgery to see how this compares with the other combination.
  Other Names: Palonosetron; Saline Solution
  Arms: Palonosetron only
Drug: Palonosetron with Dexamethasone — Women/Men 18-55 scheduled for surgery 1-3 hours in duration will be given .075 mg IV Palonosetron (Aloxi) with 8mg IV Dexamethasone (Decadron) before surgery to see if this reduces PONV.
  Other Names: Palonosetron; Aloxi; Dexamethasone; Decadron
  Arms: Palonosetron with Dexamethasone

SUMMARY:
The purpose of this study is to determine if subjects who receive Palonosetron plus Dexamethasone have less post-operative nausea and vomiting (PONV) than those who receive Palonosetron alone.

DETAILED DESCRIPTION:
Post-operative nausea and vomiting (PONV) is a frequent complication of surgery, with considerable medical and economic impact. It is also associated with high levels of patient discomfort and dissatisfaction. To many patients, PONV is a distressing event that reportedly is more feared than post-operative pain. The cause of PONV is complex and can be due to multiple factors. These factors may include certain characteristics of the patient (such as female gender, non-smoking status, and having experienced PONV in the past), the surgical procedure (intra-abdominal laparoscopic procedures, gynecologic surgeries, breast surgeries), and the type of anesthetic that is used. Untreated, the incidence of post-operative nausea and vomiting (PONV) in high risk patients can reach 70-80%. In addition, it is important to note that PONV can present during the first 24 hours after surgery or beyond. PONV alone is one of the leading causes for delayed discharge and unplanned hospital admission following outpatient surgery. Furthermore, more than 35% of surgical outpatients experience PONV following discharge, many of whom did not experience nausea or vomiting in the recovery room.

An important factor in the development of Post-operative nausea and vomiting (PONV) appears to be the release of the biogenic amine serotonin (5-HT3) in the brainstem and the peripheral nervous system. Serotonin induces nausea and vomiting via the 5-HT3 receptor.

Currently, medications that block the 5-HT3 receptor are widely accepted as a first-line anti-emetic in both the prevention and treatment of PONV. Ondansetron is the most commonly prescribed. An intra-venous dose of Ondansetron administered intra-operatively is predicted to reduce PONV by 15-20% when compared to patients who receive a placebo. However, Ondansetron has a half-life of approximately six hours and must be re-dosed in patients with prolonged or delayed-onset PONV.

By contrast, Palonosetron is another 5-HT3 receptor antagonist that has a longer half-life than Ondansetron, thus reducing the need for re-dosing; a single dose of Palonosetron was shown to be superior to a single dose of Ondansetron in the treatment of delayed nausea and vomiting associated with chemotherapy.

Furthermore, there is now evidence that a multimodal approach to the prevention of post-operative nausea and vomiting is more effective than any single medication. A recent study determined that a combination regimen of Ondansetron and Dexamethasone (a steroid medication known to prevent nausea and vomiting) provided significantly better prophylaxis against PONV than Ondansetron alone.

Therefore, the rationale for conducting this study is to evaluate whether the administration of a single dose of Palonosetron combined with Dexamethasone is superior to a single dose of Palonosetron alone in the prevention of both immediate and delayed PONV in high risk patients undergoing laparoscopic abdominal or gynecologic surgery.

In order to answer the question of whether Palonosetron plus Dexamethasone is significantly more effective at reducing the incidence of PONV than Palonosetron alone, we will enroll patients that are high risk for PONV who are undergoing laparoscopic abdominal or gynecologic surgery. This subset includes: female patients, non-smokers, and patients with a history of PONV.

Each study patient will receive Palonosetron alone or Palonosetron plus Dexamethasone immediately prior to the start of her/his surgery. We will then use an 11 point nausea scale to determine how many patients had a complete response to the medication (complete response = NO nausea and NO vomiting at any time during the study period of 0-72 hours post surgery). If a patient does experience nausea or vomiting, we will record the time and severity of the PONV as well as whether any medication was given to relieve the nausea and vomiting. If a patient is discharged from the hospital before their 72nd hour post surgery, (s)he will receive a journal in which to record any symptoms or nausea or vomiting and a member of the research team will call to obtain the information.

We predict that the combination of Palonosetron plus Dexamethasone will be superior to Palonosetron alone in the prevention of PONV. We will compare the incidence of patients with a complete response to the study medication (NO nausea and NO vomiting for 72 hours post surgery) to determine if this hypothesis is valid.

ELIGIBILITY:
Inclusion Criteria:

* Has signed an informed consent form
* Have an American Society of Anesthesiologists (ASA) Physical Status Classification of I, II, or III
* Female, 18-55 years old

  * surgically sterilized, or
  * pre-menopausal, with a negative pregnancy test within 7 days before study medication administration
* Male, 18-55 years old, who has more than 3 risk factors for PONV
* Undergoing outpatient laparoscopic gynecological surgery or laparoscopic abdominal surgery, scheduled for between 1 and 3 hours duration
* Known to have a history of post-operative nausea and vomiting and/or a history of motion sickness
* Has been a non-smoker for at least the previous 12 consecutive months
* Is able and willing to complete a subject diary until the end of the 96 Hour Follow-Up Assessment period
* Will be available to respond to follow-up by study personnel at 72 and 96 hours post emergence from anesthesia

Exclusion Criteria:

* Has an ASA Physical Status Classification of IV or V
* Is pregnant or breastfeeding
* Has been taking more than 10-15mg of oxycodone, or an equivalent opioid dose, on a regular, daily basis, for more than 3 consecutive days before surgery
* Has received an investigational drug in the precious 30 days or who is schedule to receive any investigational drug during the study period
* Has persistent or recurrent nausea and/or vomiting due to other etiologies, including but not limited to, gastric outlet obstruction, hypercalcemia, active peptic ulcer, increased intracranial pressure, or brain metastases
* Experienced retching or vomiting or uncontrolled nausea within 48 hours before administration of study drug
* Received medication with known or potential antiemetic activity within 24 hours before receiving study drug. This includes, but is not limited to: phenothiazines, butyrophenones, hydroxyzine, lorazepam, cannabinoids, metoclopramide, corticosteroids (with the exception of topical steroids for skin disorder and inhaled steroids for respiratory disorders), trimethobenzamide, monoamine oxidase inhibitors, lithium, and 5-HT3 receptor antagonists. Subjects who might require one or more of these medications during the 24-hour treatment period, other than as described in this protocol, are also excluded.

  * Note: benzodiazepines other than lorazepam are allowed within 24 hours before and during study period, but only when used for indications such as anxiety or to induce sleep.
* Received radiation therapy to abdomen or pelvis in the 7 days prior to receiving study medication and/or will receive radiation therapy to abdomen or pelvis in the evaluation period.
* Has a history of poorly controlled diabetes mellitus
* Has a history of wound dehiscence
* Has had an incidence of necrotizing fasciitis, or any similar infectious process, within the previous 90 days
* Has a know systemic fungal infection, history of tuberculosis, or other mycobacterial infection
* Is immunocompromised - defined as a white blood cell (WBC) count of <3,000 mm3
* Has any current or past medical condition (e.g., vagotomy) and/or require medication to treat a condition that could confound the evaluation of the data collected in this clinical trail
* Has a known hypersensitivity or contraindication to palonosetron hydrochloride or any another 5-HT3 receptor antagonist, dexamethasone, or any scheduled anesthetic or analgesic agents
* Has a known hypersensitivity to fentanyl and/or ketorolac tromethamine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanna Blitz, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

REFERENCES:
- [Result] Blitz JD, Haile M, Kline R, Franco L, Didehvar S, Pachter HL, Newman E, Bekker A. A randomized double blind study to evaluate efficacy of palonosetron with dexamethasone versus palonosetron alone for prevention of postoperative and postdischarge nausea and vomiting in subjects undergoing laparoscopic surgeries with high emetogenic risk. Am J Ther. 2012 Sep;19(5):324-9. doi: 10.1097/MJT.0b013e318209dff1. PMID 21519222
- See also: pubmed abstract — http://www.ncbi.nlm.nih.gov/pubmed/21519222

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from July 2010 until December 2011 in pre-surgical clinic and in same day surgery.
Groups:
- Palonosetron With Placebo: Women/Men 18-55 scheduled for surgery 1-3 hours in duration will be given .075 mg IV Intravenous Palonosetron and Saline solution
Period: Overall Study
Arm/Group | Palonosetron With Dexamethasone | Palonosetron With Placebo
Started | 59 | 59
Completed | 59 | 59
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Palonosetron With Dexamethasone | Palonosetron Only | Total
Number analyzed (Participants) | 59 | 59 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 59 | 118
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (8.8) | 36.2 (8.1) | 35.7 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 52 | 100
  Male | 11 | 7 | 18
Region of Enrollment [Number; unit: participants]
  United States | 59 | 59 | 118

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: A Complete Response (CR): defined as no nausea, no vomiting/retching, no rescue medication and no withdrawal of consent from the time of administration of the study drug(s) until 72 hours post emergence from anesthesia.
Time Frame: Pre-op through 72 hours post emergence from anesthesia
Measure: Number; unit: participants
Arm/Group | Palonosetron With Dexamethasone | Palonosetron Only
Number analyzed (Participants) | 59 | 59
participants
  0-2 Hours - no rescue medication | 38 | 38
  0-6 Hours - no rescue medication | 32 | 32
  0-72 Hours - no rescue medication | 32 | 26

2. Secondary Outcome: Number of Participants Who Experienced no or Reduced Post-Operative Nausea Vomiting (PONV) the First 96 Hours After Surgery
Description: Participants with no or reduced post operative nausea over a 96 hour period after surgery. questionnaires answered after surgery at 2 hour, 6 hour, 12 hour 72 hour and 96 hours post surgery.
Time Frame: Pre-op through 96 hours post-op
Measure: Number; unit: participants
Groups:
- Dexamethasone: Women/Men 18-55 scheduled for surgery 1-3 hours in duration will be given .075 mg IV Palonosetron (Aloxi) with 8mg IV Dexamethasone (Decadron) before surgery.
- Placebo: Women/Men 18-55 scheduled for surgery 1-3 hours in duration will be given .075 mg IV Intravenous Palonosetron and Saline solution
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 59 | 59
participants | 32 | 26

ADVERSE EVENTS:
Time Frame: We looked for adverse events from the PACU to 72 hours after surgery
Arm/Group | Palonosetron With Dexamethasone | Palonosetron Only
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 0/59 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No